CLINICAL TRIAL: NCT06619210
Title: A Multicenter, Randomized, Placebo and Active Controlled, Phase II Clinical Study to Evaluate the Efficacy and Safety of HL231 Solution for Inhalation in Patients with Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Trial to Evaluate the Safety and Efficacy of HL231 Solution for Inhalation in Patients with COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HEISCO-231-201
Record Dates: First submitted 2024-09-12; First posted 2024-10-01 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- HL231 Dose 1（Part A） (Experimental): single dose, oral inhalation by PARI BOY nebulizer
  Interventions: Drug: HL231 Dose 1/2/3/4
- HL231 Dose 2（Part A） (Experimental): single dose, oral inhalation by PARI BOY nebulizer
  Interventions: Drug: HL231 Dose 1/2/3/4
- HL231 Dose 3（Part A） (Experimental): single dose, oral inhalation by PARI BOY nebulizer
  Interventions: Drug: HL231 Dose 1/2/3/4
- Ultibro （Part A） (Active Comparator): Ultibro capsule for inhalation, consisting of a fixed dose combination of indacaterol 110µg and glycopyrronium 50µg, single dose, oral inhalation by Breezhaler
  Interventions: Drug: HL231 Dose 1/2/3/4
- Placebo Solution for Inhalation (Part A) (Placebo Comparator): Placebo Solution for Inhalation, single dose, oral inhalation by PARI BOY nebulizer
  Interventions: Drug: HL231 Dose 1/2/3/4
- HL231 Dose 2（Part B） (Experimental): single dose, oral inhalation by PARI BOY nebulizer
  Interventions: Drug: HL231 Dose 1/2/3/4
- HL231 Dose 4（Part B） (Experimental): single dose, oral inhalation by PARI BOY nebulizer
  Interventions: Drug: HL231 Dose 1/2/3/4
- Active Comparator （Part B） (Active Comparator): Ultibro capsule for inhalation, consisting of a fixed dose combination of indacaterol 110µg and glycopyrronium 50µg, single dose, oral inhalation by Breezhaler
  Interventions: Drug: HL231 Dose 1/2/3/4

INTERVENTIONS:
Drug: HL231 Dose 1/2/3/4 — HL231 Solution for Inhalation, dose 1/2/3 (Part A) , dose 2/4（Part B） single dose, oral inhalation by PARI BOY nebulizer

SUMMARY:
To evaluate the efficacy and safety of HL231 Solution for Inhalation vs Ultibro in Chinese patients with moderate to severe COPD.

DETAILED DESCRIPTION:
This study is a randomized, single-dose, multi-center, two-part, crossover, dose-ranging study of HL231 in the treatment of subjects with COPD. This study is divided into 2 parts.

Part A is a 5 treatment period single dose study. Each treatment period will be separated by a washout period of at least 14 days. The primary comparison for bronchodilation was between HL231 doses vs Ultibro or placebo in COPD patients.

Part B is a 3 treatment period single dose study. Each treatment period will be separated by a washout period of at least 14 days. The primary comparison for pharmacokinetic profile was between HL231 vs Ultibro in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of Chinese ethnicity, at least 40 years of age;
* Patients with with a clinical diagnosis of moderate to severe COPD confirmed by spirometry according to according to GOLD criteria；
* Current or ex-smokers with a>10 year pack history；
* Patients with a post-bronchodilator Forced Expiratory Volume in one second (FEV1) < 80% and ≥ 30% of the predicted normal value , and post-bronchodilator FEV1/FVC (Forced Vital Capacity) < 0.70 at visit 1；
* Patients have airway reversibility based a ≥12% increase in FEV1 following ipratropium and salbutamol treatment；
* Patients on no maintenance/background therapy or could withhold prohibited COPD medications in protocol during the screening and treatment period (except study-supplied salbutamol as an rescue medication);
* Modified Medical Research Council (mMRC) grade of at least 2 at visit 1.

Exclusion Criteria:

* Patients with any of the following significant diseases: α-1 antitrypsin deficiency, cystic fibrosis, significant asthma, active bronchiectasis, obliterated bronchiolitis, active pulmonary tuberculosis, sarcoidosis, lung fibrosis, pulmonary hypertension, pulmonary edema, interstitial lung disorder, lung cancer or other active pulmonary disease；
* Evidence or history of other clinically significant cardiovascular disease or abnormality (such as, but not limited to, unstable ischemic heart disease, congestive heart failure, uncontrolled hypertension, uncontrolled coronary artery disease, myocardial infarction, arrhythmia, long QT syndrome, paroxysmal atrial fibrillation), renal, neurological, endocrine, immunological, psychiatric, gastrointestinal, hepatic, or hematological disease or abnormality which, in the opinion of the investigator, would put the patient at risk through study participation, or would affect the study analyses if the disease exacerbates during the study;
* Patients with paradoxical bronchospasm, narrow-angle glaucoma, symptomatic benign prostatic hyperplasia(benign prostatic hyperplasia patients who were stable on treatment could have been considered), bladder-neck obstruction, severe renal impairment, or urinary retention, or any other medical history, which, in the opinion of the investigator, would contraindicate the use of an anticholinergic agent;
* Hospitalization for COPD or pneumonia within 12 weeks prior to screening (Visit 1) or screening;
* Patients who have had a COPD exacerbation that required treatment with antibiotics, systemic steroids , hospitalization or emergency treatment in the 12 weeks prior to screening (Visit 1);
* Patients who have had an acute (viral or bacterial) upper or lower respiratory tract infection, sinusitis, pharyngitis or urinary tract infections within 6 weeks prior to screening (Visit 1) or screening;
* Patients with conditions contraindicated for treatment with or having a history of allergy or hypersensitivity to any of the following inhaled drugs, drugs of a similar class or any component thereof: Anticholinergic/muscarinic receptor antagonist, Long- or short-acting β2-agonists, Sympathomimetic amines, Lactose/milk proteins, or any of the other excipients of the delivery system;
* History of frequent COPD exacerbations of moderate to severe severity averaging 2 or more per year, over the last 3 years.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2023-05-29 (Actual); Study Completion 2023-05-29 (Actual)

PRIMARY OUTCOMES:
Part A：Change from baseline in Forced Expiratory Volume in 1 Second Area Under the Curve (FEV1 AUC) 0-12 Hours | Up to 12 hours after investigational product administration
Part B：Pharmacokinetic variables: AUC0-t | Up to 144 hours after investigational product administration
Part B：Pharmacokinetic variables: AUC0-∞ | Up to 144 hours after investigational product administration
Part B：Pharmacokinetic variables: Cmax | Up to 144 hours after investigational product administration

SECONDARY OUTCOMES:
Part A & Part B：Change from baseline in Forced Expiratory Volume in 1 Second Area Under the Curve (FEV1 AUC) 0-24 Hours | Up to 24 hours after investigational product administration
Part A & Part B：Change from baseline in Forced Expiratory Volume in 1 Second Area Under the Curve (FEV1 AUC) 0-4 Hours | Up to 4 hours after investigational product administration
Part B：Change from baseline in Forced Expiratory Volume in 1 Second Area Under the Curve (FEV1 AUC) 0-12 Hours | Up to 12 hours after investigational product administration
Part B: Pharmacokinetic variables: Tmax | Up to 144 hours after investigational product administration
Part B: Pharmacokinetic variables: t1/2 | Up to 144 hours after investigational product administration
Part A & Part B：Adverse event rate | From the time of informed consent up to 14 (±2) days after the last dose of investigational product.
  Adverse events are summarized according to the system organ classification and standard name, and the system organ classification and standard name are arranged in descending order of the frequency of the tested preparation group

CONTACTS AND LOCATIONS:
Overall Officials: Zhu Luo, M.D., Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu Q, Zhao L, Yang G, Wen F, Xie L, Xiao Z, Chen F, He Q, Bian T, Xiong H, Li F, Yue Y, Li Y, Luo L, Luo Z. Efficacy, pharmacokinetics, and safety of nebulized HL231 inhalation solution in patients with chronic obstructive pulmonary disease: a randomized trial. J Thorac Dis. 2025 Oct 31;17(10):7459-7472. doi: 10.21037/jtd-2025-1130. Epub 2025 Oct 9. PMID 41229760